CLINICAL TRIAL: NCT01010607
Title: Use of Tendon Vibration and Mirror for the Improvement of Upper Limb Function and Pain Reduction After Stroke
Brief Title: Use of Tendon Vibration and Mirror for the Improvement of Upper Limb Function and Pain Reduction
Acronym: VibMirror
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Elior Moreh/ MD, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0305-09-HMO-CTIL
Record Dates: First submitted 2009-11-08; First posted 2009-11-10 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2009-11

CONDITIONS: Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Vibraton Mirror (VM) (Experimental): subjects will receive tendon vibration AND mirror therapy
  Interventions: Device: Vibration and Mirror
- Mirror (M) (Active Comparator): Subjects will receive treatment only with Mirror, together with sham vibration (over bone instead of tendon)
  Interventions: Device: Mirror therapy
- Sham (S) (Sham Comparator): Opaque board instead of mirror, bone vibration instead of tendon vibration
  Interventions: Device: no mirror, sham vibration

INTERVENTIONS:
Device: Vibration and Mirror — 10 treatments of 30 minutes in which vibration of 50-100 Hz will be administrated to the elbow and wrist muscles together with the use of a mirror. The patient moves his healthy hand in a certain repetitive pattern and watches its reflection on a mirror. Meanwhile he receives vibration in his affected hand in a timing that induces the illusion of movements similar to the movements of his healthy hand, thereby inducing a strong illusion of movement of his affected hand.
  Arms: Vibraton Mirror (VM)
Device: Mirror therapy — 10 sessions of mirror therapy: moving the healthy hand while watching its reflection on a mirror. Meanwhile sham vibration over bone in the affected handwill be given to resemble the conditions of the experimental arm.
  Arms: Mirror (M)
Device: no mirror, sham vibration — 10 sessions in which patient moves his healthy hand and tries to move his affected hand, which is hidden by an opaque board instead of a mirror. Sham vibration is applied to bone instead of muscle, no illusion is generated.
  Arms: Sham (S)

SUMMARY:
Upper limb paralysis following stroke is a very common problem. Only 30% of stroke patients who suffer from upper limb paresis experience a full recovery of function. There is a need for the development of more efficient rehabilitation methods for the improvement of the paralysed upper limb function.

It has been shown that the use of mirror therapy after a stroke induces the activation of motor, sensory and associative regions in the affected hemisphere and is associated with an improvement in the function of the affected limb. Mirror therapy is a treatment modality in which the affected arm is hidden from the patient's sight; the patient is instructed to watch the reflection of his healthy hand on a mirror while he performs movements with his healthy hand and tries to move simultaneously his affected hand. This induces the illusion that his affected hand moves well.

It has also been shown that applying vibration to a muscle tendon at frequencies between 50-100 Hz induces an illusion of elongation of the vibrated muscle, if visual feedback is prevented. For instance, vibrating the triceps will induce a strong illusion of elbow flexion.

In the present study the investigators will couple the use of a mirror with the application of vibration to tendons, in order to obtain a multisensorial and strong illusion of movement in the paralyzed limb.

The study hypothesis is that the administration of mirror therapy together with vibration will induce the activation of multiple motor, sensory and associative areas in the affected brain hemisphere, resulting in improvement of the affected upper limb function, compared to the administration of mirror therapy alone or sham therapy.

ELIGIBILITY:
Inclusion Criteria:

* Stroke onset 1 month-1 year ago
* NIH Stroke Scale 3-15 on admission to study
* Affected Upper limb function 10-90% on Fugl-Meyer scale
* Ability to understand instructions and to move freely the unaffected upper limb

Exclusion Criteria:

* Severe cognitive impairment- severe Aphasia or severe Neglect that impair ability to understand instructions or to execute tasks

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-12 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Upper Limb function according to Fugl-Meyer assessment | after treatment, and 3 months after treatment

SECONDARY OUTCOMES:
Activity of Daily living performance assessed by FIM (Functional Independence Measurement) score | after treatment and 3 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel

REFERENCES:
- [Background] Goodwin GM, McCloskey DI, Matthews PB. The contribution of muscle afferents to kinaesthesia shown by vibration induced illusions of movement and by the effects of paralysing joint afferents. Brain. 1972;95(4):705-48. doi: 10.1093/brain/95.4.705. No abstract available. PMID 4265060
- [Result] Dohle C, Pullen J, Nakaten A, Kust J, Rietz C, Karbe H. Mirror therapy promotes recovery from severe hemiparesis: a randomized controlled trial. Neurorehabil Neural Repair. 2009 Mar-Apr;23(3):209-17. doi: 10.1177/1545968308324786. Epub 2008 Dec 12. PMID 19074686